CLINICAL TRIAL: NCT06242691
Title: A Phase 1/2 Open-label Study to Evaluate the Safety and Efficacy of MK-1200 in Participants With Advanced Solid Tumors
Brief Title: Safety and Efficacy of MK-1200 in Participants With Advanced Solid Tumors (MK-1200-002)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1200-002; 2023-508684-68-00 (Registry Identifier: EU CT); U1111-1298-7820 (Registry Identifier: UTN); MK-1200-002 (Other: MSD)
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Antiemetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: MK-1200 (Experimental): In Part 1, participants will receive escalating doses of MK-1200 via intravenous (IV) infusion every 2 weeks (Q2W) until any discontinuation criteria are met.
  Interventions: Biological: MK-1200; Drug: Antiemetic
- Part 2: MK-1200 Cohort A (Experimental): In Part 2, participants in Cohort A will receive either Dose 1 or Dose 2 of MK-1200 via IV infusion Q2W until any discontinuation criteria are met.
  Interventions: Biological: MK-1200; Drug: Antiemetic
- Part 2: MK-1200 Cohort B (Experimental): In Part 2, participants in Cohort B will receive Dose 1 of MK-1200 via IV infusion Q2W until any discontinuation criteria are met.
  Interventions: Biological: MK-1200; Drug: Antiemetic

INTERVENTIONS:
Biological: MK-1200 — IV Infusion
Drug: Antiemetic — One or more prophylactic antiemetic(s) (e.g. 5-HT3 receptor antagonists, dexamethasone, neurokinin-1 receptor antagonists, etc.) may be selected based on previous response of participants to antiemetic medications and individual factors, and will be administered per approved product label prior to MK-1200 infusion

SUMMARY:
The purpose of this study is to assess the efficacy and safety of MK-1200 monotherapy in participants with advanced/metastatic gastric/gastroesophageal junction (GEJ) cancer, esophageal cancer, biliary tract cancer, and pancreatic ductal adenocarcinoma who have received, or been intolerant to, all treatments known to confer clinical benefit. Part 1 of the study will be a dose escalation to determine the maximum tolerated dose (MTD). Part 2 will evaluate safety and efficacy of MK-1200 at 2 different doses

ELIGIBILITY:
Inclusion Criteria:

* Confirmed advanced (unresectable and/or metastatic) solid tumor: gastric cancer (including gastroesophageal junction cancer), esophageal cancer, biliary tract cancer, or pancreatic ductal adenocarcinoma
* Participants who experienced Adverse Events (AEs) due to previous anticancer therapies must have recovered to < Grade 1 or baseline
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy
* Hepatitis B surface antigen (HBsAg) positive participants are eligible if they have received Hepatitis B Virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load
* Participants with a history of Hepatitis C Virus (HCV) infection are eligible if HCV viral load is undetectable
* Received and progressed on or after 1 or 2 prior lines of therapy

Exclusion Criteria:

* Active severe digestive disease
* History of acute myocardial infarction; unstable angina; stroke or transient ischemic attack within 6 months prior to the first dose of study intervention
* Diabetes or hypertension that cannot be controlled by medication
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Received prior systemic anticancer therapy including investigational agents within 4 weeks before study intervention
* Received prior radiotherapy within 2 weeks of start of study intervention, or has radiation-related toxicities, requiring corticosteroids
* Known additional malignancy that is progressing or has required active treatment within the past 2 years
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Active infection requiring systemic therapy
* Have not adequately recovered from major surgery or have ongoing surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants who Experience One or More Dose-Limiting Toxicities (DLTs) | Up to approximately 28 days
  The occurrence of any of the following toxicities within 28 days after the first dose of study intervention will be considered a DLT, if assessed by the investigator to be possibly, probably, or definitely related to study intervention administration:
  * Grade 4 nonhematologic toxicity (not laboratory). Any nonhematologic AE ≥Grade 3 in severity should be considered a DLT, with pre-specified exceptions
  * Any Grade 3 or Grade 4 laboratory value (hematologic or nonhematologic), with pre-specified exceptions
  * Febrile neutropenia Grade 3 or Grade 4 as prespecified by the protocol
  * Prolonged delay (>2 weeks) in initiating Cycle 2 due to intervention-related toxicity
  * Any intervention-related toxicity that causes the participant to discontinue intervention during Cycle 1
  * Missing >25% of MK-1200 doses as a result of drug-related AEs during the first cycle
  * Grade 5 toxicity
Number of Participants who Experience One or More Adverse Events (AEs) | Up to approximately 16 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported for each arm.
Number of Participants who Discontinue Study Intervention Due to an AE | Up to approximately 15 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study intervention due to an AE will be reported for each arm.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1) as assessed by Blinded Independent Central Review (BICR) | Up to approximately 16 months
  ORR is defined as the percentage of participants who have achieved confirmed Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by blinded independent central review (BICR).
ORR per RECIST 1.1 as Assessed by Investigator | Up to approximately 16 months
  ORR is defined as the percentage of participants who have achieved confirmed Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by the investigator.
Area under the curve (AUC) of MK-1200 | Cycles 1 and 4: predose and 0.5, 2, 4, 8, 24, 48, 96, 168, and 240 hours postdose; Cycles 2-3 Days 1 and 8: predose and 0.5 hours postdose; Day 1 of Cycles 5 onward (up to 15 months): predose and 0.5 hours postdose. Cycle is 14 days.
  AUC is defined as the area under the concentration versus time curve. Blood samples will be collected at pre-specified timepoints to determine AUC.
Minimum Concentration (Cmin) of MK-1200 | Cycles 1 and 4: predose and 0.5, 2, 4, 8, 24, 48, 96, 168, and 240 hours postdose; Cycles 2-3 Days 1 and 8: predose and 0.5 hours postdose; Day 1 of Cycles 5 onward (up to 15 months): predose and 0.5 hours postdose. Cycle is 14 days.
  Cmin is defined as the minimum concentration of MK-1200 observed in plasma after its administration and just prior to administration of a subsequent dose. Blood samples will be collected at pre-specified timepoints to determine Cmin.
Maximum Concentration (Cmax) of MK-1200 | Cycles 1 and 4: predose and 0.5, 2, 4, 8, 24, 48, 96, 168, and 240 hours postdose; Cycles 2-3 Days 1 and 8: predose and 0.5 hours postdose; Day 1 of Cycles 5 onward (up to 15 months): predose and 0.5 hours postdose. Cycle is 14 days.
  Cmax is defined as the maximum or 'peak' concentration of MK-1200 observed after its administration. Blood samples will be collected at pre-specified timepoints to determine Cmax.
Duration of Response (DOR) per RECIST 1.1 as Assessed by BICR | Up to approximately 16 months
  For participants demonstrating a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from the first documented evidence of a CR or a PR until Progressive Disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. The DOR as assessed by BICR will be reported.
DOR per RECIST 1.1 as Assessed by Investigator | Up to approximately 16 months
  For participants demonstrating a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from the first documented evidence of a CR or a PR until PD or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. The DOR as assessed by the investigator will be reported.
Progression-Free Survival (PFS) per RECIST 1.1 as Assessed by BICR | Up to approximately 16 months
  PFS is defined as the time from randomization to the first documented PD by BICR or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR will be reported.
PFS per RECIST 1.1 as Assessed by Investigator | Up to approximately 16 months
  PFS is defined as the time from randomization to the first documented PD by investigator or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by the investigator will be reported.
Overall Survival (OS) | Up to approximately 16 months
  OS is defined as the time from randomization to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (16):
- United States (5):
  - The University of Louisville, James Graham Brown Cancer Center ( Site 0004), Louisville, Kentucky
  - START Midwest ( Site 0014), Grand Rapids, Michigan
  - South Texas Accelerated Research Therapeutics (START) ( Site 0005), San Antonio, Texas
  - START Mountain Region ( Site 0015), West Valley City, Utah
  - University of Virginia Health System-Hematology-Oncology ( Site 0009), Charlottesville, Virginia
- The Alfred Hospital ( Site 0103), Melbourne, Victoria, Australia
- Bradfordhill-Clinical Area ( Site 0301), Santiago, Region M. de Santiago, Chile
- China (3):
  - Beijing Cancer hospital-Digestive Oncology ( Site 0401), Beijing, Beijing Municipality
  - Fujian Cancer Hospital-oncology department ( Site 0409), Fuzhou, Fujian
  - First Huai'an Hospital Affiliated to Nanjing Medical University ( Site 0415), Huai'an, Jiangsu
- Israel (5):
  - Rambam Health Care Campus-Oncology Division ( Site 0602), Haifa
  - Hadassah Medical Center ( Site 0604), Jerusalem
  - Rabin Medical Center-Oncology ( Site 0603), Petah Tikva
  - Sheba Medical Center ( Site 0605), Ramat Gan
  - Sourasky Medical Center ( Site 0601), Tel Aviv
- Samsung Medical Center-Division of Hematology/Oncology ( Site 1003), Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26319&tenant=MT_MSD_9011